CLINICAL TRIAL: NCT05135754
Title: Investigation of Patient Benefits With a New Supporting Ostomy Product and Support Service in Patients With a Newly Stoma Formation
Brief Title: Investigation of Patient Benefits With a New Supporting Ostomy Product in Patients With a Newly Stoma Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP340
Record Dates: First submitted 2021-10-27; First posted 2021-11-26 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-04

CONDITIONS: Stoma Ileostomy; Stoma Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test product - new supporting ostomy product and support service (Other): The arm includes the newly developed supporting ostomy product (leakage notification system Heylo) used together with a support service
  Interventions: Device: Heylo

INTERVENTIONS:
Device: Heylo — Test of the supporting product (test product) for a 12 weeks period. No additional intervention will be conducted. A few follow up nurse calls to assess few endpoints together with subject. All remaining endpoints are captured via surveys send to the subjects every 14 days.

SUMMARY:
People with intestinal stomas can have, despite development of better ostomy products, problems with leakage which influence their quality of life negatively.

To overcome this, Coloplast has developed a new supporting ostomy product called Heylo™, which has an adhesive sensor layer that should be placed underneath the baseplate. The sensor layer consists of an electronic sensor system that continuously detects moisture and output leakage underneath the baseplate. A transmitter connected to the sensor layer continuously evaluates the incoming information and sends a status to a smartphone software application, which based on a predefined flow decides which information to deliver to the user about the baseplate status.

ELIGIBILITY:
Inclusion Criteria:

1. Have provide written informed consent.
2. Be at least 18 years of age and have full capacity.
3. Have had their stoma for less than 9 months.
4. Have intact skin on the peristomal area (assessed by investigator)
5. Be able to use one of the five test products (i.e. Ø40, Ø50, Ø60, Ø70, Ø80 mm)
6. Ileo- or colostomists with liquid and/or mushy output (Bristol scale type 5-7)
7. Is willing to refrain from use of paste and protective sheets.
8. Have a smartphone applicable for the HeyloTM app.
9. Have been self-managing stoma appliance for at least 14 days.
10. Are able to follow study procedures for 3 months (assessed by investigator)
11. Are willing to receive their ostomy products through Coloplast Charter for the duration of the study.

Exclusion Criteria:

1. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
2. Is breastfeeding.
3. Is pregnant based on urine pregnancy test.
4. Enrolled in another current research study or have previously participated in this investigation.
5. Has known hypersensitivity towards any of the products used in the investigation.
6. Is using/have a pacemaker.
7. Has a complicated stoma at baseline (dehiscence/prolapse/hernia)
8. Has limited life expectancy or receive palliative care.
9. Has stage 4 cancer.
10. Having more than one stoma synchronously
11. Having ongoing non-healed abdominal wounds
12. Reoperation / stoma reversal planned during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brady, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (10):
- United Kingdom (10):
  - Southmead/North Bristol NHS Trust, Bristol
  - Chelsea & Westminster Hospital, Chelsea
  - Devon/Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Norfolk/James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Leeds/Leeds Teaching Hospitals NHS Trust, Leeds
  - Illingworth, Manchester
  - Middlesbrough/South Tees NHS trust, James Cook University Hospital, Middlesbrough
  - Newcastle University/The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Petersborough/ North West Anglia NHS Foundation trust, Petersborough City Hospital, Peterborough
  - Preston/Lancashire Teaching Hospitals NHS Trust, Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brady RR, Sheard D, Alty M, Vestergaard M, Boisen EB, Ainsworth R, Hansen HD, Ajslev TA. Novel digital leakage notification system can promote better stoma management routines: a multicentre clinical trial. Br J Nurs. 2025 Jan 13;34(1):14-22. doi: 10.12968/bjon.2025.0278. PMID 39792106
- [Derived] Brady RRW, Sheard D, Alty M, Vestergaard M, Boisen EB, Ainsworth R, Hansen HD, Ajslev TA. Evaluating the Effect of a Novel Digital Ostomy Device on Leakage Incidents, Quality of Life, Mental Well-Being, and Patient Self-Care: An Interventional, Multicentre Clinical Trial. J Clin Med. 2024 Sep 24;13(19):5673. doi: 10.3390/jcm13195673. PMID 39407731

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product - New Supporting Ostomy Product and Support Service: The arm includes the newly developed ostomy support product together with a support service
  Heylo: Test of the supporting product (test product) for a 12 weeks period. No measurement will be conducted. All endpoints are captured via surveys send to the subjects every 14 days.
Period: Overall Study
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Started | 100 (Safety population)
Baseline (Intention to Treat Population) | 92
Completed | 80
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 92
Age, Continuous [Mean (Full Range); unit: years] | 49.4 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Times With Stoma Effluent Leakage Outside the Baseplate (e.g. Onto Clothes or Bedsheets) Within the Last 2 Weeks
Description: Survey question: Think back on the last 2 weeks; how many times have you experienced stoma effluent leakage outside the baseplate (e.g. onto clothes or bedsheets)?
Time Frame: Baseline (Day 0) and Final Evaluation (Week 12)
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of leakages per two weeks
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 92
Number of leakages per two weeks
  Baseline | 1.57 [1.19 to 2.08]
  Final evaluation | 0.93 [0.56 to 1.54]
Statistical Analysis 1: Comparison: Test Product - New Supporting Ostomy Product and Support Service; Test type: Superiority; p = 0.046, Mixed Models Analysis; Risk Ratio (RR) = 0.59, 95% CI 2-sided [0.35 to 0.99]

2. Secondary Outcome: Patient Self-management
Description: Patient Activation Measure (PAM) score The Patient Activation Measurement (PAM) is scored on a scale ranging from 0 to 100.
  Individuals who score high on this instrument typically understand the importance of taking a pro-active role in managing their health and have the skills and confidence to do so.
Time Frame: Baseline (Day 0) and Final Evaluation (Week 12)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 92
score on a scale
  Baseline | 68.201 [64.677 to 71.726]
  Final evaluation | 74.815 [71.217 to 78.414]
Statistical Analysis 1: Comparison: Test Product - New Supporting Ostomy Product and Support Service; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 6.61, 95% CI 2-sided [3.45 to 9.78]

3. Secondary Outcome: Ostomy Leakage Impact Tool - 'Emotional Impact' Domain
Description: Leakage-related quality of life. The Ostomy Leakage Impact (OLI) tool consists of 22 item questions, which are grouped in three domains. The three domains concern the impact of stoma leakage on (1) 'emotional' aspects, (2) 'usual and social activities', and (3) 'coping and in control'. Each domain has a score ranging from 0-100. A score of 100 equals no impact and a score of 0 represents full negative impact, thus a higher score means that subjects are less impacted from leakage in their daily life.
Time Frame: Baseline (Day 0) and Final Evaluation (Week 12)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 92
score on a scale
  Baseline | 57.124 [52.375 to 61.873]
  Final evaluation | 77.136 [72.280 to 81.991]
Statistical Analysis 1: Comparison: Test Product - New Supporting Ostomy Product and Support Service; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 20.01, 95% CI 2-sided [15.02 to 25.00]

4. Secondary Outcome: Ostomy Leakage Impact Tool - 'Usual and Social Activities' Domain
Description: as for outcome 3
Time Frame: Baseline (Day 0) and Final Evaluation (Week 12)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 90
score on a scale
  Baseline | 82.750 [78.447 to 87.054]
  Final Evaluation | 89.072 [84.726 to 93.418]
Statistical Analysis 1: Comparison: Test Product - New Supporting Ostomy Product and Support Service; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 6.32, 95% CI 2-sided [2.71 to 9.94]

5. Secondary Outcome: Ostomy Leakage Impact Tool - 'Coping and in Control' Domain
Description: as for outcome 3
Time Frame: Baseline (Day 0) and Final Evaluation (Week 12)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 92
score on a scale
  Baseline | 62.779 [57.586 to 67.973]
  Final Evaluation | 77.082 [71.757 to 82.408]
Statistical Analysis 1: Comparison: Test Product - New Supporting Ostomy Product and Support Service; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 14.30, 95% CI 2-sided [8.26 to 20.35]

6. Secondary Outcome: Health Related Quality of Life
Description: The EQ-5D-5L instrument consists of five dimensions with five predetermined levels of response that is used to generate a health state profile, which then can be assigned a summary index score. Translation of health states and index scores are based on the specific value set for United Kingdom.
  The index scores based on the value set for United Kingdom ranges from -0.285 to 1.
  Index score of -0.285 is the worst health state. Index score of 1 is the best health state.
Time Frame: Baseline (Day 0) and Final Evaluation (Week 12)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 92
score on a scale
  Baseline | 0.713 [0.663 to 0.763]
  Final evaluation | 0.747 [0.696 to 0.798]
Statistical Analysis 1: Comparison: Test Product - New Supporting Ostomy Product and Support Service; Test type: Superiority; p = 0.075, Mixed Models Analysis; Mean Difference (Final Values) = 0.03

7. Secondary Outcome: EQ-5D-5L Visual Analogue Scale (VAS)
Description: Subjects rate their perceived health from 0 (worst imaginable health) to 100 (best imaginable health).
Time Frame: Baseline (Day 0) and Final Evaluation (Week 12)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Test Product - New Supporting Ostomy Product and Support Service
Number analyzed (Participants) | 92
score on a scale
  Baseline | 71.771 [68.089 to 75.453]
  Final evaluation | 76.454 [72.713 to 80.196]
Statistical Analysis 1: Comparison: Test Product - New Supporting Ostomy Product and Support Service; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 4.68, 95% CI 2-sided [1.55 to 7.81]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the study period being 12 weeks ± 2 weeks.
Groups:
- Safety Population: n=100 subjects were recruited for the study. All n=100 subjects were included as the safety population. Eight subjects were omitted from the ITT population, as they had not used the Test Product. Six of the eight subjects were screening failures, a single subject wished to discontinue, and a single subject was lost to follow-up before the first visit (V1; baseline).
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 5/100
Other Adverse Events (participants affected / at risk) | 20/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=100)
Patient was admitted into the hospital for subarachnoid hemorrhage and encephalitis (Nervous system disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Low Neutrophils (Blood and lymphatic system disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Bleeding Stoma (Gastrointestinal disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Diarrhoea (Gastrointestinal disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Vomiting (Gastrointestinal disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Admitted to hospital as a result for producing high output black stoma contents (Gastrointestinal disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Intestinal Blockage (Gastrointestinal disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
Intestinal infection (Gastrointestinal disorders) | 1 (1) — Not related to Test Product (Assessed by investigators)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=100)
Skin redness and irritation (Skin and subcutaneous tissue disorders) | 18 (20) — Assessed by investigators to be possibly, probably, or causally related to the Test Product
Headache (Nervous system disorders) | 6 (7) — Not related to Test Product; Not related to Procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05135754/Prot_SAP_000.pdf